#### **DURABILITY PAS**

The US Study for Evaluating Endovascular Treatments of Lesions in the Superficial Femoral Artery and Proximal Popliteal By using the Everflex Nitinol Stent System Post Approval Study

Statistical Analysis Plan Version 2.0 26 September 2018

NCT01680835




| Medtronic<br>Statistical Analysis Plan | |
|---|---|
| Clinical Investigation Plan Title | The US StuDy for EvalUating EndovasculaR TreAtments of Lesions in the Superficial Femoral Artery and Proximal Popliteal By usIng the EverfLex NitInol STent System Post Approval Study DURABILITY PAS |
| Clinical Investigation Plan Identifier | CP-1001 |
| Clinical Investigation Plan Version | Version 3.1 |
| Sponsor | Medtronic<br>3033 Campus Drive Suite N550<br>Plymouth, MN 55441 |
| Document Version | Version 2.0; 26-Sep-2018 |

Revision [2.0]

#### **Confidentiality Statement**

The information contained in this document is confidential and the proprietary property of Medtronic. Any distribution, copying, or disclosure without the prior written authorization of Medtronic is strictly prohibited. Persons to whom the information is disclosed must know that it is confidential and that it may not be further disclosed by them.

Form

Revision [2.0]




## **Table of Contents**

| 1. | ' | Version History | 3 |
|----|-----|--------------------------------------------------|---|
| 2. | ı | List of Abbreviations and Definitions of Terms | 3 |
| 3. | | Introduction | 3 |
| 4. | : | Study Objectives | 3 |
| 5. | | Investigation Plan | 5 |
| 6. | I | Determination of Sample Size | 5 |
| | Pri | imary Endpoint and Sample Size Adjustment | 5 |
| | Jus | stification of Performance Goal | 5 |
| | Po | tential Outcomes | 6 |
| | Saı | mple Size and Power | 7 |
| 7. | : | Statistical Methods | 8 |
| | 7.1 | 1 Study Subjects | 8 |
| | 7.2 | 2 General Methodology | 9 |
| | 7.3 | 3 Center Pooling | 9 |
| | 7.4 | 4 Handling of Missing Data and Dropouts | 9 |
| | 7.5 | 5 Demographic and Other Baseline Characteristics | 9 |
| | 7.6 | 5 Treatment Characteristics | 0 |
| | 7.7 | 7 Evaluation of Objectives | 0 |
| | 7.8 | 8 Safety Evaluation | 0 |
| | 7.9 | 9 Changes to Planned Analysis1 | 0 |
| 8. | , | Validation Requirements | 0 |
| 9. | | References | 2 |

Revision [2.0]




#### 1. Version History

| Version | Summary of Changes | Author(s)/Title |
|---|---|---|
| 1.0 | Not Applicable, New Document | , Principal Statistician |
| 2.0 | <ul> <li>Updated this SAP to reflect the new SOP template and Protocol Version 3.1. Added Section 4 Study Objectives, Section % Investigation Plan, Section 6</li> <li>Determination of Sample Size, Section 7 Statistical Methods and Section 9</li> <li>Reference.</li> </ul> | , Principal Statistician |

#### 2. List of Abbreviations and Definitions of Terms

| Abbreviation | Definition |
|--------------|---------------------------------|
| AE | Adverse Event |
| CIP | Clinical Investigation Plan |
| PG | Performance Goal |
| SAP | Statistical Analysis Plan |
| TLR | Target Lesion Revascularization |
| TVR | Target Vessel Revascularization |

#### 3. Introduction

This document outlines the detailed statistical methods to be implemented for the data collected within the scope of the Medtronic Durability PAS Study. The purpose of this plan is to provide a framework within which answers to the study objectives can be achieved in a statistically rigorous fashion, without bias or analytical deficiencies. Specifically, this Plan has the following purpose: To prospectively (a priori) outline the types of analyses and presentations of data that will form the basis for conclusions to be reached that will answer the clinical evaluation objectives outlined in the protocol, and to explain in detail how the data will be handled and analyzed, adhering to commonly accepted standards and practices of biostatistical analysis in the medical device industry. Results obtained from the analyses outlined in this document will be the basis of the Final Study Report for the overall Clinical Investigational Plan (CIP).

## 4. Study Objectives

The purpose of this study is to confirm the safety and effectiveness of primary stenting with the EverFlex™ Self-Expanding Peripheral Stent System (EverFlex stent) when used in subjects with atherosclerotic stenoses, restenoses or occlusions of the native superficial femoral artery or superficial femoral and proximal popliteal arteries through three years post-procedure.

Revision [2.0]




**Primary Endpoint:** The primary endpoint of the study is composite endpoint defined as freedom from acute death, freedom from 36-month amputation, and freedom from 36-month clinically-driven target lesion revascularization compared to a PTA performance goal.

#### **Secondary Endpoints:**

- **1. Freedom from Stent Fracture:** Determined by x-ray at 1, 2 and 3 years using the following classifications:
  - Class 0 No strut fractures
  - Class I Single tine fracture
  - Class II Multiple tine fractures
  - Class III Stent fracture(s) with preserved alignment of the components
  - o Class IV Stent fracture(s) with mal-alignment of the components
  - o Class V Stent fracture(s) in a trans-axial spiral configuration

#### AND the following categories:

- Category A − Restenosis ≤ 50% at site of fracture
- Category B Restenosis > 50% at site of fracture
- Category C Occlusion at site of fracture
- Category D Unable to determine
- 2. Freedom from acute death, freedom from amputation and freedom from clinically-driven target lesion revascularization at 1 and 2 years: Defined as the absence of all-cause mortality occurring within 30-days, absence of any major amputation within 12-/24- months and the absence of any clinically-driven repeat invasive procedure, including angioplasty, stenting, endarterectomy, bypass, or thrombolysis, performed to open or increase the lumen diameter inside or within 10 mm of the previously treated lesion due to the return of clinical symptoms within 12-/24-months of the procedure.
- **3. Freedom from 36-month amputation:** Defined as the absence of any major amputation (removal of the target limb or a part of the target limb above the metatarsal line) within 36 months of the procedure.
- **4. Freedom from 36-month clinically-driven target lesion revascularization:** Defined as the absence of any clinically-driven repeat invasive procedure, including angioplasty, stenting, endarterectomy, bypass, or thrombolysis, performed to open or increase the lumen diameter inside or within 10 mm of the previously treated lesion due to the return of clinical symptoms within 36 months of the procedure.
- **5. Freedom from acute death:** Defined as the absence of all-cause mortality occurring within 30-days of the procedure.
- **6. Device Success:** Defined as the ability to deploy the stent as intended at the treatment site.

# [DPAS] Statistical Analysis Plan Revision [2.0]  Medtronic

- 7. Improvement in Rutherford Clinical Category at 1 Year: Defined as an improvement in clinical status indicated by a decrease of one or more in Rutherford Clinical Category compared to baseline.
- **8. Improvement in Ankle-Brachial Index at 1 Year:** Defined as an increase in the ankle-brachial index (ABI) compared to baseline in subjects with compressible arteries and baseline ABI < 0.9.
- 9. Walking Improvement at 1 Year: Defined as an increase in Walking Impairment Questionnaire score in subjects who did not have iliac disease treated at the time of the index procedure compared to baseline.
- **10. Adverse Event Rate:** Defined as the rate of adverse events that occur during the course of the study; event and subject counts as well as proportions of subjects with events categorized by type will be reported. Note that adverse events are captured at each study assessment. Counts and rates of all-cause mortality will be reported both as part of the overall adverse event profile as above, and separately as a specific outcome.

#### 5. Investigation Plan

DURABILITY PAS is a prospective, multi-center, non-randomized, single arm study with sequential enrollment of all qualified subjects undergoing treatment of atherosclerotic lesions in the native superficial femoral artery or the superficial femoral and proximal popliteal arteries. All eligible subjects who provide informed consent will undergo PTA and stenting using the EverFlex device. Follow-up will take place at pre-discharge, 30 days, 1 year, 2 years and 3 years.

## 6. Determination of Sample Size

#### **Primary Endpoint and Sample Size Adjustment**

The study's primary endpoint has been previously defined. The associated statistical hypothesis is that the resulting event-free rate at 36 months is greater than the Performance Goal (PG), which is adapted from RESILIENT 3-year data on freedom from TLR for PTA subjects.

The null and alternative hypotheses for the primary endpoint are:

 $H_0$ :  $\pi_t \le \pi_{pg}$   $H_a$ :  $\pi_t > \pi_{pg}$ 

where  $\pi_t$  is the event-free rate in subjects treated with an EverFlex device and  $\pi_{pq}$  is the PG of 35%.

Analysis of this endpoint will be carried out by Kaplan-Meier methods. The point estimate of the event-free rate at 36 months (1095 days) from the date of the index procedure will be computed along with its one-sided 97.5% lower confidence bound. If the lower bound is greater than 35%, it will be declared that the PG and the corresponding primary study objective have been met.

#### **Justification of Performance Goal**

The structure of the composite endpoint is derived from a 12-month composite endpoint described by VIVA Physicians Inc. (VPI) as part of their development of safety and effectiveness Performance Goals (PG) for the use of bare nitinol stents in the treatment of femoropopliteal lesions.<sup>1, 2</sup> The VPI 12-month



composite was defined as acute death, index limb amputation and target vessel revascularization (TVR) through 12-months. This composite event rate in the studies reviewed was 30.5% at 12 months (Table 1). However, there were no long-term follow-up to 3 years reported.

**Table 1: PTA Performance Goals - Safety Data** 

| | Company A | Company B | Company C | Combined |
|---|---|---|---|---|
| | (n=29) | (n=24) | (n=63) | (n=116) |
| 12 month Composite<br>(acute death, 12m<br>TVR, 12m amputation | 38.5% (10/26) | 33.3% (6/18) | 25.5% (13/51) | 30.5% (20/95) |

Three-year data on freedom from TLR was presented on the PTA arm of the RESILIENT study.<sup>3</sup> The reported event-free rate at 3 years among RESILIENT subjects randomized to PTA treatment was 41.8%, a value which is adjusted as follows to account for longer lesions enrolled in DURABILITY II.

The statistical model employed is a Cox regression on the outcome of freedom from TLR applied to DURABILITY II data. Lesion length (in mm) as measured by the core laboratory was the predictor of outcome, resulting in a point estimate of 0.01543 for the logarithm of the hazard ratio, and therefore a hazard ratio of  $e^{0.01543}$ =1.0155 per mm of lesion length (with longer lesions associated with lower freedom-from-TLR rates).

As the mean lesion length in RESILIENT was 68 mm versus 89 mm in DURABILITY II, the resulting adjusted event-free rate can be obtained using a formula analogous to adjusting with odds ratios:

$$\pi_{pg}/(1-\pi_{pg}) = (0.418/(1-0.418))*1.0155^{(89-68)}$$

Solving this equation gives  $\pi_{pg}$  = 0.342, which is rounded up to give the PG of 35%. Note that this PG is conservative in that it (1) does not attempt to account for any other systematic differences between RESILIENT and DURABILITY II and (2) does not explicitly account for the other elements of the composite endpoint (since these were not presented for RESILIENT), which if included would lower the expected freedom-from-event rate below that seen for TLR alone.

#### **Potential Outcomes**

Table 2 summarizes approximate outcomes under potential results for freedom from event, using binomial estimation. Note that the actual analysis will be conducted using time-to-event methods and is subject to currently unknown censoring times, and that therefore the actual success criteria will vary slightly from those noted below.




| Table 2: Approxima | Table 2: Approximation to Possible Outcomes and Corresponding 97.5% Lower Confidence Bound <b>Primary Endpoint (PG=35%)</b> | | |
|---|---|---|---|
| Sample Size | Count of subjects with freedom from event | 36-Month Freedom From<br>Event Rate | 97.5% lower<br>confidence bound |
| 108 | 48 | 44.4% | 35.1% |
| 108 | 49 | 45.4% | 36.0% |
| 108 | 50 | 46.3% | 36.9% |
| 108 | 51 | 47.2% | 37.8% |

Revision [2.0]

#### Sample Size and Power

The required sample size for evaluating the primary endpoint can be approximated using the normal method for testing a single proportion (as above, under Kaplan-Meier methods the actual power will vary slightly from this calculation):

$$n = \frac{(\pi_{pg} \times (1 - \pi_{pg})) \times (Z_{1 - \alpha} + Z_{1 - \beta} \sqrt{\pi_{t} (1 - \pi_{t}) / (\pi_{pg} (1 - \pi_{pg})))^{2}}}{(\pi_{t} - \pi_{pg})^{2}}$$

Where,

- Type I error (α) = 0.025 (one-sided)
- Statistical power  $(1 \beta) = 90\%$
- Z is the standard normal deviate for  $\alpha$  =0.025 and  $\beta$ =0.10.
- $\pi_t$  is estimated freedom-from-event at 36 months
- $\pi_{pg}$  is the PG

Using this approximation with  $\pi_t$  = 0.55 (estimated from current DURABILITY II data),  $\pi_{pg}$  = 0.35 (the *a priori* performance goal),  $Z_{1-\alpha}$  = 1.96 and  $Z_{1-\beta}$  = 1.28 gives a sample size of 62. Allowing for approximately 30% of subjects lacking a 3-year follow-up visit, the needed sample size under this approximation for 90% power is a minimum of 89.

An additional sample size requirement is based on the secondary endpoint of freedom from stent fracture at 1 year. In DURABILITY I and DURABILITY II, 1-year stent fracture rates of 8.1% (n=151) and 0.4% (n=287), respectively, were observed. The pooled fracture rate of these two studies is 3.0% (13/438), around which a confidence interval of specified width is desired. The desired precision is 7.2%

Revision [2.0]




(half-width of 3.6%); we therefore find a 95% two-sided normal confidence interval with upper bound 3.0% + 3.6% = 6.6%, and extract the relevant sample size.

**Table 3: Sample Size Freedom from Stent Fracture** 

| | Sample Size for Freedom from Stent Fracture | | |
|---|---|---|---|
| Sample Size | Count of subjects with event | Event Rate | 97.5% upper<br>confidence bound<br>(95% two-sided) |
| 95 | 3 | 3.16% | 6.67% |
| 96 | 3 | 3.13% | 6.61% |
| 97 | 3 | 3.09% | 6.54% |
| 98 | 3 | 3.06% | 6.47% |

From the above table, the required sample size at 1 year is 97 subjects. Considering a 10% rate of attrition, a minimum of 108 subjects are needed, which is larger than the sample size of 89 calculated for the primary endpoint. The enrolled sample size is therefore 108. Please note that multiple stents are allowed in each subject in the study. The stent fracture endpoint will be analyzed on stent level. To be conservative, sample size calculation is performed on subject level. Therefore, more stents than the above assumption may be included in the analysis.

#### 7. Statistical Methods

## 7.1 Study Subjects

#### 7.1.1 Disposition of Subjects

The number of subjects who are selected, and who have a scheduled follow-up visit will be summarized at each scheduled visit.

#### 7.1.2 Clinical Investigation Plan (CIP) Deviations

Protocol deviations will be reported descriptively by counts of type and listing by site.

#### 7.1.3 Analysis Sets

All study subjects with non-missing values will be included in the primary endpoint analysis and secondary endpoint analysis.

#### 7.2 General Methodology

All statistical analyses will be performed using Statistical Analysis System (SAS) for Windows (version 9.2 or above, SAS Institute Inc. Cary, N.C.) or other widely accepted statistical or graphical software. In general, data for all study subjects combined will be presented. Individual data will be presented in subject listings.

Descriptive statistics will be used to present the data and to summarize the results. Discrete variables will be presented using frequency distributions and cross-tabulations. Continuous variables will be summarized by presenting the number of observations (N), mean, standard deviation, median, minimum, and maximum values.

For adverse event reporting, the primary analysis will be based on subject counts, not event counts. A subject with more than one event will be counted only once toward the event rate based on the total number of subjects with adverse events.

Unless otherwise specified, statistical significance will be declared when p<0.05 for two-sided tests and p<0.025 for one-sided tests such as the primary endpoint.

#### 7.3 Center Pooling

This is a multi-center clinical study, with standardization of subject enrollment, data entry and adverse event reporting. All investigational sites will follow the requirements of a common protocol, data collection procedures and case report forms. To present the data from this clinical study in a summary form, a comparison across all sites will be completed to determine if the generated data could be pooled. The following variables will be completed to assess the appropriateness of pooling data from across all sites:

- Baseline demographics such as age and gender
- Lesion characteristics such as lesion length and percent stenosis

The distributions of the above variables across the sites will be tabulated.

## 7.4 Handling of Missing Data and Dropouts

In general, imputation of missing data will not be performed for all analyses. Subjects who dropped out will be censored at date of last follow-up contact.

## 7.5 Demographic and Other Baseline Characteristics

All demographic, medical history and clinically relevant baseline variables will be summarized and tabulated. Descriptive statistics will be presented as follows:

 Categorical variables, including binary variables, will be reported by giving the number and percentage of patients in each category.



• Continuous variable will be reported by presenting the number of observations, mean, standard deviation, median, IQR, minimum, and maximum of each variable

#### 7.6 Treatment Characteristics

Device success defined as the ability to deploy the stent as intended at the treatment site will be reported.

### 7.7 Evaluation of Objectives

Analysis of the primary endpoint will be carried out by Kaplan-Meier methods. The point estimate of the event-free rate at 36 months (1095 days) from the date of the index procedure will be computed along with its one-sided 97.5% lower confidence bound. If the lower bound is greater than 35%, it will be declared that the PG and the corresponding primary study objective have been met.

For secondary endpoints, descriptive statistics will be provided. No formal statistical hypothesis testing will be performed. Categorical variables will be analyzed using frequency tabulation and event rate. For continuous variables, analysis will include mean, median, standard deviation, and ranges. Time-to-event variables including the primary endpoint and the secondary endpoint of freedom from stent fracture will be analyzed using survival analysis and reported at 1 year (365 days), 2 years (730 days) and 3 years (1095 days), with Kaplan-Meier plots provided.

#### 7.8 Safety Evaluation

All Adverse Events (AEs) will be coded using pre-specified AE Code in the CEC charter. The AEs will be adjudicated by CEC. Frequencies and percentages of AEs will be presented.

## 7.9 Changes to Planned Analysis

There is no change to the planned analysis. Any changes to planned statistical analyses determined necessary prior to performing the analyses will be documented in an amended Statistical Analysis Plan and approved prior to the analysis. Any other deviations or changes from the planned analyses deemed necessary due to violation of critical underlying statistical assumptions, data characteristics, or missing data will be clearly described in the clinical study report with justification and rationale.

## 8. Validation Requirements

| | Objectives | Validation level (Level I;<br>Level II) |
|------------------|------------|-----------------------------------------|
| Primary Endpoint | | |

Revision [2.0]




| | Objectives | Validation level (Level I;<br>Level II) |
|---|---|---|
| | Composite endpoint defined as freedom from acute death, freedom from 36-month amputation, and freedom from 36-month clinically-driven target lesion revascularization compared to a PTA performance goal. | Dataset = Level I, Graph=Level II |
| Secondary<br>Endpoints | | |
| | 1.Freedom from Stent Fracture | Dataset = Level I,<br>Graph=Level II |
| | 2. Freedom from acute death, freedom from amputation and freedom from clinically driven target lesion revascularization at 1 and 2 years | Dataset = Level I, Graph=Level II |
| | 3. Freedom from 36-month amputation | Dataset = Level I,<br>Graph=Level II |
| | 4. Freedom from 36-month clinically-driven target lesion revascularization | Dataset = Level I,<br>Graph=Level II |
| | 5. Freedom from acute death | Dataset = Level I, Graph=Level II |
| | 6. Device Success | Level I |
| | 7. Improvement in Rutherford Clinical<br>Category at 1 Year | Level I |
| | 8. Improvement in Ankle-Brachial Index at 1 Year | Level I |
| | 9. Walking Improvement at 1 Year | Level I |

Medtronic 

**Form** 

Revision [2.0]

| | Objectives | Validation level (Level I;<br>Level II) |
|---|---|---|
| | 10. Adverse Event Rates | Dataset = Level I, |
| | | Table=Level II |
| Baseline | | |
| Demographic and | | |
| Lesion | | |
| Characteristic | | |
| | Baseline Demographic and Lesion | Dataset = Level I, |
| | Characteristic | Table=Level II |
| Follow up<br>Compliance | | |
| Comphanice | Follow up compliance | Dataset = Level I, |
| | Tonow up compliance | Table=Level II |
| <b>Protocol Deviation</b> | | |
| | Protocol Deviations | Dataset = Level I, |
| | | Table=Level II |

#### 9. References

- 1. Rocha-Singh KJ. Proposed Performance Goals for Single-Arm Clinical Trials of Bare Nitinol Stents in the Femoral Popliteal Artery. Vascular InterVentional Advances. Las Vegas, NV2006.
- Rocha-Singh KJ, Jaff MR, Crabtree TR, Bloch DA, Ansel G. Performance goals and endpoint 2. assessments for clinical trials of femoropopliteal bare nitinol stents in patients with symptomatic peripheral arterial disease. Catheter Cardiovasc Interv. May 1 2007;69(6):910-919.
- 3. Katzen B. Long-Term RESILIENT Data for Nitinol Stenting in the SFA. Vascular Interventional Advances (VIVA). Las Vegas2011.